CLINICAL TRIAL: NCT00704132
Title: A Randomized, Placebo-Controlled Study to Evaluate the Safety, Efficacy and Mechanism of Action of MK0431/Sitagliptin in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Brief Title: Sitagliptin Mechanism of Action Study in Patients With Type 2 Diabetes Mellitus (0431-059)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0431-059; 2006_511
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Results first posted 2011-05-16 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- sitagliptin (Experimental): Participants randomized to this arm will be administered sitagliptin 100mg daily, for six weeks.
  Interventions: Drug: Comparator: sitagliptin phosphate
- Placebo (Placebo Comparator): Participants randomized to this arm will be administered matching placebo, daily for six weeks.
  Interventions: Drug: Comparator: placebo (unspecified)

INTERVENTIONS:
Drug: Comparator: sitagliptin phosphate — Sitagliptin tablet 100 mg, administered once daily before the morning meal.
  Arms: sitagliptin
Drug: Comparator: placebo (unspecified) — Matching placebo tablet, administered once daily before the morning meal.
  Arms: Placebo

SUMMARY:
A clinical study to determine the safety, efficacy and the way sitagliptin works in patients with Type 2 Diabetes Mellitus who have inadequate glycemic (blood sugar) control.

ELIGIBILITY:
Inclusion Criteria:

* Participant has type 2 diabetes mellitus
* Males
* Females who are highly unlikely to become pregnant
* Participants poorly controlled without taking any, or taking one or two oral antidiabetic medications

Exclusion Criteria:

* Participant has a history of type 1 diabetes mellitus or history of ketoacidosis
* Participant required insulin therapy within the prior 8 weeks
* Participant is on or has been taking TZDs such as Actos® (pioglitazone) or Avandia® (rosiglitazone) within the prior 12 weeks of the screening visit

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-02-14 (Actual); Primary Completion 2010-04-28 (Actual); Study Completion 2010-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Muscelli E, Casolaro A, Gastaldelli A, Mari A, Seghieri G, Astiarraga B, Chen Y, Alba M, Holst J, Ferrannini E. Mechanisms for the antihyperglycemic effect of sitagliptin in patients with type 2 diabetes. J Clin Endocrinol Metab. 2012 Aug;97(8):2818-26. doi: 10.1210/jc.2012-1205. Epub 2012 Jun 8. PMID 22685234

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 57 participants were enrolled in this study. Of these, 7 participants with normal fasting glucose (NFG) only underwent pre-randomization experiments and did not receive an allocation number, were not randomized to one of the treatment groups, and did not receive double-blind study medication.
Groups:
- Sitagliptin: Participants were administered sitagliptin 100 mg tablet once daily before the morning meal for six weeks.
- Placebo: Participants were administered sitagliptin matching placebo tablet once daily before the morning meal for six weeks.
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 26 | 24
Completed | 25 | 22
Not Completed | 1 | 2
Not completed — Clinical Adverse Experience | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Customized [Number; unit: participants] | 26 | 24 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 19 | 16 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glucose 5-Hour Incremental AUC at Week 6
Description: Participants underwent the 5-hour meal test prior to randomization (baseline) and was repeated at the conclusion of the 6-week double-blind study period. The change from baseline in Glucose 5-Hour Incremental AUC at Week 6 is computed as the difference between the Week 6 measurement and the baseline measurement.
Time Frame: Baseline and Week 6
Population: Full-Analysis-Set (FAS) population, which includes all randomized participants who had a baseline value, received at least one dose of randomized treatment, and had a measurement at Week 6.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg*hr/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 25 | 22
mg*hr/dL | -83.9 (87.7) [-125.9 to -41.9] | 27.0 (84.3) [-16.0 to 70.1]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in Least-Squares Mean = -111.0, 95% CI [-158.0 to -63.9] — Sitagliptin minus Placebo

ADVERSE EVENTS:
Description: The analyses for all safety outcomes used the All Patients as Treated (APaT) approach. The APaT population used all randomized participants who received at least 1 dose of study therapy.
Arm/Group | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=26) | Placebo (N=24)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.